CLINICAL TRIAL: NCT06538870
Title: Dental Implant Healing in Patients Taking Tumor Necrosis Factor (TNF)-Alpha Inhibitors
Brief Title: Dental Implant Healing With TNF-Alpha Inhibitors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Nobel Biocare (Industry)
Responsible Party: Principal Investigator, Katherine France, Assistant Professor of Oral Medicine, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1778 SA France
Record Dates: First submitted 2024-07-24; First posted 2024-08-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Edentulism; Dental Implants; TNF-alpha Inhibitors
Keywords: Dental implants; TNF-alpha inhibitors; Biologic agents; Missing teeth
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Intervention Model Description: Two groups will be recruited, one taking TNF-alpha inhibitors and one not taking these medications but matched via age and sex to the first group. Both will receive dental implant placement to replace missing teeth and both will be followed at the same intervals, using the same outcome measures, and for the same length of time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients taking TNF-alpha inhibitors (Experimental): Adult patients (18 years of age or older) taking a TNF-alpha inhibitor as defined by the NIH and missing teeth will be recruited to receive dental implant placement according to standard of care for ideal dental restoration. Patients must have been taking a stable dose of the drug for at least 6 months and have no contra-indications to implant placement (regular tobacco use in the last year, periodontal disease, pathology in the jaw bone(s), history of head and neck radiation, history of antiresorptive or antiangiogenic agents, uncontrolled diabetes, pregnancy, other medical conditions that preclude safe delivery of outpatient medical care) to be eligible for enrollment in the study.
  Interventions: Procedure: Placement of dental implants
- Patients not taking TNF-alpha inhibitors (Experimental): Patients over age 18 not taking TNF alpha inhibitors will be recruited and matched via age and sex to the patients taking TNF-alpha inhibitors. The general exclusion criteria (regular tobacco use in the last year, periodontal disease, pathology in the jaw bone(s), history of head and neck radiation, history of antiresorptive or antiangiogenic agents, uncontrolled diabetes, pregnancy, other medical conditions that preclude safe delivery of outpatient medical care) will apply to both arms equally.
  Interventions: Procedure: Placement of dental implants

INTERVENTIONS:
Procedure: Placement of dental implants — Dental implants will be placed in the edentulous area as per standard surgical procedure and as appropriate to bring the patient to standard of care restoratively.

SUMMARY:
The goal of this pilot study is to learn about healing after dental implant placement in patients taking a class of biologic drug called Tumor Necrosis Factor or TNF-alpha antagonist or inhibitor. The main questions it aims to answer are:

Do patients taking TNF-alpha inhibitors have any complications after the placement of dental implants? Do patients taking TNF-alpha inhibitor experience increased pain after dental implant placement compared to the expected levels when healing from this procedure? Researchers will recruit patients both taking these drugs and those not taking these drugs to compare the outcomes between the two groups.

Participants missing teeth will be recruited to receive dental implants to meet ideal dental status and will be followed before and after the implant placement to determine levels of health and ensure proper healing. Participants will be followed for a total of one year and follow up visits will consist of both clinical examination and radiographs (x-rays) to evaluate bone level and implant status. Participants will also be asked to rate their pain during clinic visits and at home on a diary and record the amount of pain control medication they take after the implant procedure.

DETAILED DESCRIPTION:
This descriptive study will recruit 15 patients requiring implant restoration as standard of care for missing teeth taking a stable dose (unchanged for 6 months or more) of a TNF-α inhibitor, regardless of the targeted disease and 15 patients requiring implant restoration not taking TNF-alpha inhibitors (30 patients total). Patients will be recruited without age restrictions or limitations on systemic medical conditions or other medications, although patients not taking TNF-alpha inhibitors will be matched via age and sex to those taking the medications. Patients with periodontal disease and smokers will not be included given the known connection between these comorbidities and compromised implant outcomes. Patients will be selected based on inclusion and exclusion criteria, consent, availability, and willingness to follow study protocols. Patients will not stop their TNF-alpha or any other medication during the study period to minimize adverse systemic outcomes.

Once enrolled, subjects will be evaluated according to medical history including reason for TNF inhibitor, demographics, and clinical and radiographic features. NobelParallel conical connection implants will be placed under standard surgical approach to confirm equanimity of experience. Nobel anatomical healing abutments will be placed above each implant and followed for 12 months according to study procedures. All patients will receive the same dental implants, specifically the NobelParallel TiUltra 3.75x11.5 implant and titanium healing abutment (see product guide attached).

Follow up appointments will assess healing including pain score and analgesic use (routine standard of care but will be recorded as part of this research study), periodontal probing, and radiographs. Radiographs will determine bone quality and quantity. Nature and frequency have been planned according to best practices, with details found below. The images proposed that are additional to routine clinical care are: CBCT immediately after implant placement, CBCT at 6 months following implant placement, periapical radiographs at 6 and 12 months after implant placement. Patient serum will be drawn at the implant placement and all follow up visits to test for complete blood count, C-reactive protein, and erythrocyte sedimentation rate to assess systemic inflammation and any changes after surgery. If patients complete all study visits, their implant placement surgical treatment will be financially covered in full. Patients will also be compensated for their time during the 3,6, and 12 month study visits, which will improve patient retention. Of these, the 3 month study visit would be routine during normal clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Require placement of implants to assist with dental restoration.
* Half of the patients (15) will be recruited with the key criteria of a TNF-alpha inhibitor medication that they have been taking consistently without dose adjustment or other changes for at least 6 months. The other half will be recruited without a target medical condition but will be recruited to match the patients taking TNF-alpha inhibitors in age and gender.
* All patients will be medically fit to withstand implant placement as judged by best practice applied by the study team.
* The patients will be required to read and speak English
* All patients must either provide their own independent consent for medical procedures or to attend study visits with a surrogate decision maker.

Exclusion Criteria:

Patients will not be excluded on the basis of age (within the adult population), race, economic status, sex or gender, or other demographic factors. Patients will be excluded if:

* They have periodontal disease (periodontal pockets above 4mm in the applicable arch or radiographic evidence of horizontal bone loss more than mild severity)
* There is other evidence of pathology in the treated arch on pre-treatment review including radiographs, such as any evidence of cyst or tumor formation in the mandible.
* They have uncontrolled diabetes (HbA1c >8.0) as confirmed by evaluating labs taken on anyone with diagnosed diabetes in the 6 months before the study enrollment.
* They have history of head and neck radiation for any reason
* They are taking any antiresorptive or antiangiogenic agents for any reason including osteoporosis, multiple myeloma, bone metastasis of other primary cancers
* They are unable to seek outpatient medical care or are not medically fit to withstand implant placement, including those with critical findings or lab values. Medical exclusion of patients will be completed by the investigators based on standard of care for surgical procedures in dental medicine and based on specific implant guidelines.
* Patients who have routinely used tobacco or tobacco products in the last 1 year will be excluded, as tobacco use is a known contributor to poor prognosis after implant placement. For this reason, dental implant placement is only recommended in patients who have quit or never used tobacco products.

  * Pregnant women are unlikely to meet inclusion criteria as dental implant placement is considered an elective procedure and typically deferred in dentistry until after delivery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety of implant placement in patients taking TNF-α inhibitors | Healing will be assessed over 1 year after implant placement
  A pilot cohort of patients will be recruited who require implants for standard of care restoration for tooth loss. Patients will be evaluated pre- and post-operatively and followed for 1 year to assess healing using clinical exam.

SECONDARY OUTCOMES:
Patient pain after implant placement in patients receiving TNF-alpha inhibitors using patient rating scales | This will be assessed during the pre-surgical appointment to understand patient baseline and after surgery daily for the first week and then at 1 week, 1,3,6,and 12 months.
  While no previous dental research has directly evaluated perception of healing in patients taking TNF-α inhibitors, previous evidence points to an increase in pain during surgical healing in patients taking BAs. Patient discomfort will be measured by visual analog (VAS) patient rating scales as are widely used after dental surgery. The VAS scale from 0 to 10 where 0 means no pain and 10 means the worst possible pain will be used.
  Applying these outcomes to implant healing in patients taking TNF-α inhibitors will provide an assessment of patient experience. We hypothesize that there will be an increase in pain ratings compared to established expectations. This is the first study to evaluate patient discomfort after implant placement in patients taking BAs and the first prospective study of patients taking BAs in dental medicine and thus will add to the literature by characterizing healing and patient experience.
Patient pain after implant placement in patients receiving TNF-alpha inhibitors using analgesic use | This will be assessed during the pre-surgical appointment to understand patient baseline and after surgery daily for the first week and then at 1 week, 1,3,6,and 12 months.
  While no previous dental research has directly evaluated perception of healing in patients taking TNF-α inhibitors, previous evidence points to an increase in pain during surgical healing in patients taking BAs. Patient discomfort as measured by analgesic use in number and timing of doses taken will be evaluated. Extrapolating these outcomes to implant healing in patients taking TNF-α inhibitors will provide an assessment of patient experience. We hypothesize that there will be an increase in analgesic need compared to established expectations, to be further evaluated according to additional factors, if present, at further study. This is the first study to evaluate patient discomfort after implant placement in patients taking BAs and the first prospective study of patients taking BAs in dental medicine and thus will add to the literature by characterizing healing and patient experience.

OTHER OUTCOMES:
Systemic levels of inflammatory markers | Blood will be drawn for lab tests at implant visit and at follow up visits (1 week, 1 month, 3 month, 6 month, 12 month) to trend values.
  We will also perform exploratory analyses of whether systemic inflammation, as assessed by systemic blood markers (CRP, ESR, CBC, and cytokine measurements), is associated with implant healing, peri-implantitis, or discomfort after implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine France, DMD, MBE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD including patient outcome data will be available upon reasonable request from other researchers with similar studies, and will be shared only in aggregate and in anonymized form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 5 years after study close on reasonable request to the investigators and in aggregate form.
Access Criteria: Interested investigators may contact the study team to obtain access to the data or supporting documents.